CLINICAL TRIAL: NCT06835478
Title: Evaluate a Local Program to Reduce the Risky Use of Screens by Children Under 3, Based on the Experience of Parents Who Successfully Stopped This Exposure (EPURE)
Brief Title: Evaluate a Local Program to Reduce the Risky Use of Screens by Children Under 3, Based on the Experience of Parents Who Successfully Stopped This Exposure.
Acronym: EPURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CHSD_0032_EPURE
Record Dates: First submitted 2024-08-02; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Exposure; Child Development
Keywords: screens; screens exposure; child Development

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EPURE + (Active Comparator): In this phase, a tool will be tested aimed to reduce screen time. A screen will be conducted at 2 and 6 months to measure the program's effectiveness.
  Interventions: Behavioral: EPURE + : EPURE program
- EPURE - (Active Comparator): In this arm, no tool will be used. This arm will require only advices. Depending on the result of the screen at 2 months, adjustement will be made.
  * Failure : They will be added to the EPURE +'s arm.
  * Success : screen at 6 months
  Interventions: Behavioral: EPURE - : Standard practices

INTERVENTIONS:
Behavioral: EPURE + : EPURE program — EPURE program will be tested.
  Arms: EPURE +
Behavioral: EPURE - : Standard practices — This group will receive standard practices to prevent the use of screens in child under 3
  Arms: EPURE -

SUMMARY:
Early exposure to screens puts children at risk of later neurodevelopmental delay. This exposure is particularly prevalent among the underprivileged populations in our study area, and we don't yet know the motivations, factors and constraints that need to be put in place to remedy the situation.

Our approach is a bottom-up study, based on the experience of parents who stopped their child's exposure to screens before age 3, to develop a program to reduce early exposure to screens. This will then be tested on a larger scale via a randomized trial

DETAILED DESCRIPTION:
The research will be performed in 2 phases:

Phase 1: No intervention, an qualitative and observational phase.

We will identify participants through parents' reports during standard pediatric follow-up consultations. Those who report the cessation of screen exposure will be interviewed using the SCREEN survey, both before and at least 3 months after cessation. Our study's objectives will be presented along with an oral agreement. These "expert parents" will be contacted by phone to gather necessary data for sampling before any qualitative interview. Our aim is to have a carefully selected, homogeneous sample, rather than a representative one. Eligible parents may differ based on certain criteria, leading to potential bias : child's age, presence of older siblings, parents' socio-professional category, childcare arrangements for children <3 years of age, screen-free period (lockdown or not). Inclusion will occur after this stage.

The objectives of this interview are as follows:

1. Identify the factors that led to screen exposure.
2. Triggering factors in parents' motivation to change.
3. Practical aspects of change: obstacles, driving forces, family needs

The results of this survey will form the basis for the EPURE program. Working sessions with a multi-professional working group should define :

1. The most effective methods for transmitting information, whether visual or oral.
2. The medium used to convey the information (such as drawing, text, diagram, video, face-to-face...)
3. The chosen mode of communication, which could be vertical (conference, consultation, expert opinion) or horizontal (feedback, workshops with expert parents, etc.).
4. Proposed alternatives, such as donating or lending games, referring to socialization centers, providing psychological support, etc.

Final implementation will depend on the results of phase 1 and should not be anticipated

PHASE 2 : described as a prospective multicenter interventional study, which falls within the scope of the JARDE law.

The inappropriate use of screens will be identified by completing the SCREEN survey with all families of children under 3 years of age who attend the centers participating in the study. This identification will take place during consultations or "all-inclusive" interviews for children under 3, or during a consultation for a family member who has raised a suspicion of a high-risk situation (for example, a baby being calmed down with a cell phone during a consultation for an older child or a parent for example).

The program will involve the random selection of volunteer families in the cohort. Beforehand, a randomization list will be prepared and provided to the centers in sealed envelopes, each containing an encrypted code corresponding to the inclusion arm. This method was chosen for its minimal disruption to daily consultation practice. Neither the investigator nor the family will have access to the meaning of the code, ensuring unbiased selection.

ELIGIBILITY:
Inclusion Criteria:

* Live in Saint-Denis (France)
* Parent(s) of child(ren) for whom the family has declared that they have succeeded in stopping or totally modifying their behaviour with screens before the child's 3rd birthday (standard form for all health record follow-up examinations).
* Declaration confirmed by the negativation of the SCREEN result calculated a posteriori for two periods (before and after stopping), at least 3 months apart.
* No objection to the use of data for research purposes.

Exclusion Criteria:

* Non-French-speaking public
* Severe neurological or sensory disorder in the child
* Child in alternating custody with difficulty accessing screen exposure in the other custody arrangement.
* Refusal to use data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Demographic informationns (child) | [Day 1]
  First and last name, age
Results of SCREEN survey | [Day 1]
  SCREEN Survey's results.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hopitalier de Saint-Denis, Saint-Denis, Seine Saint Denis, France